CLINICAL TRIAL: NCT02217436
Title: iPad as a Distraction Tool During Facial Laceration Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Amy Williams, Co-Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iPadWilliams
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Anxiety; Laceration Repair; Children
MeSH Terms: conditions — Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- iPad (Experimental): iPad with age-appropriate applications, videos, and music
  Interventions: Device: iPad; Other: Standard Care
- Standard Care (Active Comparator): All study participants will receive standard care, which consists of procedural explanation and preparation by providers, verbal encouragement and comforting by providers and parents, and topical anesthetic (LET) followed by injectable lidocaine administration (whether one or both of these anesthetics will be used will be determined by the provider prior to randomization).
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: iPad — iPad with age-appropriate applications, videos, and music
  Arms: iPad
Other: Standard Care — All study participants will receive standard care, which consists of procedural explanation and preparation by providers, verbal encouragement and comforting by providers and parents, and topical anesthetic (LET) followed by injectable lidocaine administration (whether one or both of these anesthetics will be used will be determined by the provider prior to randomization).

SUMMARY:
Children aged 2-12 presenting to the Rady Children's Hospital San Diego (RCHSD) emergency department with facial lacerations requiring suture repair will be eligible to participate in the study. Participating children will be randomized to standard care versus standard care plus iPad use during the procedure. Children's anxiety levels assessed using a validated scale will be measured from video recordings made of the procedure. Parent and provider satisfaction surveys will be completed following the procedure. The primary study aim is to determine how iPad use affects children's anxiety levels during facial laceration repair. The secondary study aim is to determine how iPad use affects parent and provider satisfaction regarding a child's facial laceration repair. Hypothesis is that iPad use decreases children's anxiety levels during facial laceration repair and increases parent and provider satisfaction regarding a child's facial laceration repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patients: Male and female children aged 2-12 of all ethnic backgrounds and socioeconomic levels presenting to the emergency department for laceration repair. Children sustaining single, uncomplicated facial lacerations, which can be repaired with basic suture techniques, are eligible for the study. Lacerations repaired using LET cream, lidocaine injection, and LET cream and lidocaine injection are all eligible for the study.
2. Parents of enrolled patients.
3. Providers of enrolled patients: Residents, fellows, attendings, and nurse practitioners serving as the primary provider performing the laceration repair.

Exclusion Criteria:

1. Patients: Lacerations to parts of the body other than the face. Children with developmental disabilities. Children with laceration repair requiring sedation. Children with complex lacerations requiring subspecialty repair.
2. Parents and/or providers of children not eligible or enrolled in the study.
3. Providers: Medical students performing the laceration repair.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bema Bonsu, MD, Principal Investigator — University of California, San Diego and Rady Children's Hospital San Diego; Amy Williams, MD, Principal Investigator — University of California, San Diego and Rady Children's Hospital San Diego
Locations (1):
- Rady Children's Hospital San Diego, San Diego, California, United States

REFERENCES:
- [Background] Crellin D, Sullivan TP, Babl FE, O'Sullivan R, Hutchinson A. Analysis of the validation of existing behavioral pain and distress scales for use in the procedural setting. Paediatr Anaesth. 2007 Aug;17(8):720-33. doi: 10.1111/j.1460-9592.2007.02218.x. PMID 17596217
- [Background] Luhmann JD, Kennedy RM, Porter FL, Miller JP, Jaffe DM. A randomized clinical trial of continuous-flow nitrous oxide and midazolam for sedation of young children during laceration repair. Ann Emerg Med. 2001 Jan;37(1):20-7. doi: 10.1067/mem.2001.112003. PMID 11145766
- [Background] McQueen A, Cress C, Tothy A. Using a tablet computer during pediatric procedures: a case series and review of the "apps". Pediatr Emerg Care. 2012 Jul;28(7):712-4. doi: 10.1097/PEC.0b013e31825d24eb. PMID 22766593
- [Background] Sinha M, Christopher NC, Fenn R, Reeves L. Evaluation of nonpharmacologic methods of pain and anxiety management for laceration repair in the pediatric emergency department. Pediatrics. 2006 Apr;117(4):1162-8. doi: 10.1542/peds.2005-1100. PMID 16585311
- [Background] Jay SM, Elliott C. Behavioral observation scales for measuring children's distress: the effects of increased methodological rigor. J Consult Clin Psychol. 1984 Dec;52(6):1106-7. doi: 10.1037//0022-006x.52.6.1106. No abstract available. PMID 6520283
- [Derived] Bryl AW, Bonsu B, Johnson AL, Pommert KBJ, Hollenbach KA, Kanegaye JT. Tablet Computer as a Distraction Tool During Facial Laceration Repair: A Randomized Trial. Pediatr Emerg Care. 2021 Aug 1;37(8):e425-e430. doi: 10.1097/PEC.0000000000001626. PMID 30422942

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 eligible patients were approached and 25 refused to participate in the study (not consented), 80 participants were randomized, and 3 withdrew from the study.
Groups:
- iPad: iPad + Standard Care
  iPad: iPad with age-appropriate applications, videos, and music
  Standard Care: All study participants will receive standard care, which consists of procedural explanation and preparation by providers, verbal encouragement and comforting by providers and parents, and topical anesthetic (LET) followed by injectable lidocaine administration (whether one or both of these anesthetics will be used will be determined by the provider prior to randomization).
Period: Overall Study
Arm/Group | iPad | Standard Care
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Incomplete data | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard Care: Standard Care
  Standard Care: All study participants will receive standard care, which consists of procedural explanation and preparation by providers, verbal encouragement and comforting by providers and parents, and topical anesthetic (LET) followed by injectable lidocaine administration (whether one or both of these anesthetics will be used will be determined by the provider prior to randomization).
- Total: Total of all reporting groups
Arm/Group | iPad | Standard Care | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 38 | 77
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.0 (2.5) | 5.5 (2.6) | 5.2 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 24 | 28 | 52
Location of laceration [Count of Participants; unit: Participants]
  Forehead/eyebrow | 16 | 23 | 39
  Lip | 3 | 4 | 7
  Chin | 19 | 10 | 29
  Other | 1 | 1 | 2
Number of sutures [Mean (Standard Deviation); unit: sutures] | 4.0 (2.4) | 4.6 (2.6) | 4.3 (2.5)
Duration of procedure [Mean (Standard Deviation); unit: minutes] | 15.5 (6.5) | 16.4 (8.4) | 16.0 (7.5)
Topical anesthetic [Count of Participants; unit: Participants]
  Topical | 37 | 34 | 71
  No topical | 2 | 4 | 6
Use of restraint [Count of Participants; unit: Participants] | 20 | 19 | 39
Type of provider [Count of Participants; unit: Participants]
  Pediatric emergency medicine | 12 | 15 | 27
  Pediatrics | 8 | 5 | 13
  Emergency medicine | 2 | 2 | 4
  Nurse practitioner | 6 | 5 | 11
  Fellow | 4 | 7 | 11
  Resident | 7 | 4 | 11
Infiltrated anesthetic [Count of Participants; unit: Participants] | 30 | 30 | 60
Buffered with bicarbonate [Count of Participants; unit: Participants] | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Observational Score Behavioral Distress Revised (OSBD-R)
Description: Weighted average Observational Score Behavioral Distress Revised (OSBD-R) scored from videotapes of the entire laceration repair procedure Scale 0-23.5 (0 low/better, 23.5 high/worse)
Time Frame: Entire laceration repair procedure
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | iPad | Standard Care
Number analyzed (Participants) | 39 | 38
units on a scale | 2.3 [0 to 6.2] | 0.8 [0.1 to 5.5]
Statistical Analysis 1: Comparison: iPad vs Standard Care; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Parent Survey
Description: Parent rating of own anxiety during the procedure Likert-based scale 1-5 (1 low/better, 5 high/worse)
Time Frame: Survey administered immediately following the laceration repair
Population: Parent own anxiety survey
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | iPad | Standard Care
Number analyzed (Participants) | 39 | 38
score on a scale | 2 [1 to 4] | 4 [3.8 to 5]
Statistical Analysis 1: Comparison: iPad vs Standard Care; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | iPad | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No